CLINICAL TRIAL: NCT01984853
Title: Cardiology-Emergency Medicine Cardiac Biomarker Research Initiative
Acronym: ED~Cards
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Richard M Nowak, Principal Investigator, Henry Ford Health System
Other Study IDs: HFHS: ED-CARDS ACS Registry; HFHS: ED CARDS Registry (Registry Identifier: HFHS: ED~Cards Collaborative)
Record Dates: First submitted 2013-10-30; First posted 2013-11-15 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; repository; Observational
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — Approximately 6-8.5 ml of blood will be collected in each of two anticoagulant tube types: SST and K2EDTA plasma.
  The first blood collection in the ED is designated as t0 ED ECG time (+ 60 minutes).
  Additional blood draws of approximately 6-8.5 mL/tube type will occur at t1 = 30 (+/- 10 minutes) after t0, t2=1 (+/-15 minutes) hour after t0, t4 = 3 (+/- 15 minutes) hours after t0 (if the patient is still in the ED/hospital).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OBSERVATIONAL REGISTRY: Individuals presenting with signs and/or symptoms of Acute Coronary Syndrome at the Henry Ford Hospital Emergency Department (ED).
  Interventions: Other: OBSERVATIONAL REGISTRY

INTERVENTIONS:
Other: OBSERVATIONAL REGISTRY
  Other Names: This is an observational registry only, there are no Interventions.

SUMMARY:
This is an OBSERVATIONAL Specimen procurement and data collections trial for acute coronary syndrome that will be conducted in the Emergency Department at Henry Ford Hospital.

The standard protocol for evaluating patients in the Emergency Department for possible acute myocardial infarction includes the measurement of cardiac troponin over 3 hours. Subjects presenting to the ED with chest discomfort or ischemic symptoms will be eligible for blood draw protocol. The study is blinded to treating physicians and does not change current standard of care. After informed consent patients will have blood samples drawn at 0, 30 minutes, 1 hour and 3 hours.

Serum from the samples will be stored in a -80 research freezer to be evaluated at a later time as new cardiac markers for acute coronary syndrome are developed.

DETAILED DESCRIPTION:
Subjects considered for enrollment in this study will be identified and approached by either the Principal Investigator or trained study coordinator (SC). Candidates for enrollment will be individuals presenting with signs and/or symptoms of Acute Coronary Syndrome at the Henry Ford Hospital Emergency Department (ED).

This specimen collection study is a prospective serial draw plasma collection study designed to collect specimens for use in existing or future clinical studies. Specimen collection is expected to take approximately 30-36 months. Specimens will be collected from subjects that are being evaluated for Acute Coronary Syndrome (ACS).

Other than sample collection, no special procedures or medications are required by the study.

The study aims to enroll approximately 250-500 individuals evaluated for possible ACS in the ED.

Specimens will be obtained from the subject at the following time points:

t0 =Baseline ECG (ECG time + 60 minutes) t1= within 30 (+/- 10 minutes) minutes after t0 t2 = 1 (+/- 15 minutes) hours after t0 t3 = 3 (+/-15 minutes) hours after t0

Each sample will consist of approximately 6-8.5 ml of blood in each of two anticoagulant tube types: SST and K2EDTA plasma. Four serial specimens will be collected within 3 hours of presentation to the ED for observation of ACS.

* The Investigator or designee will obtain the subject's written informed consent prior to collecting the specimen.
* Each subject will be given a unique study number. An enrollment log will be used to document the enrollment of individuals by study number. This study number will be used to identify the individual throughout the study.
* Each subject will have a medical history reviewed and documented, as well as significant cardiac medical history documented in the subject's case report form in addition to demographic information including age, gender, race, ethnicity, and medication history.
* Each subject will have a baseline ECG obtained in the ED, vital signs and routine laboratory results. These will be documented in the subject's case report form.
* Approximately 6-8.5 ml of blood will be collected in each of two anticoagulant tube types: SST and K2EDTA plasma. The first blood collection in the ED is designated as t0 ED ECG time (+ 60 minutes). Additional blood draws of approximately 6-8.5 mL/tube type will occur at t1 = 30 (+/- 10 minutes) after t0, t2=1 (+/-15 minutes) hour after t0, t4 = 3 (+/- 15 minutes) hours after t0 (if the patient is still in the ED/hospital).
* For each draw, a minimum volume (after processing) of approximately 2 mL of plasma should be obtained. The specimens will be processed, aliquoted, and retained in a -70 secured freezer.

Inclusion/Exclusion Criteria

Inclusion Criteria:

* Patient greater than 21 years of age
* Experiencing symptoms of possible ACS
* Willing and able to comply with all aspect of the protocol

Exclusion Criteria:

* Acute distress and/or requires immediate life-saving intervention
* CPR, external defibrillation or cardioversion within 24 hours of presentation
* Unable to provide or understand the informed consent
* STEMI leading to immediate reperfusion
* Transferred from another facility
* Trauma related injuries
* Pregnancy or breast feeding

ELIGIBILITY:
Inclusion Criteria:

* Patient greater than 21 years of age
* Experiencing symptoms of possible ACS
* Willing and able to comply with all aspect of the protocol

Exclusion Criteria:

* Acute distress and/or requires immediate life-saving intervention
* CPR, external defibrillation or cardioversion within 24 hours of presentation
* Unable to provide or understand the informed consent
* STEMI leading to immediate reperfusion
* Transferred from another facility
* Trauma related injuries
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for enrollment will be individuals presenting with signs and/or symptoms of Acute Coronary Syndrome at the Henry Ford Hospital Emergency Department (ED).
Sampling Method: Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Study Objective | 4 years
  The study objective is to collect blood and plasma specimens for the assessment of ACS Biologic Assessments in patients presenting to the Emergency Department with symptoms consistent with ACS according to Henry Ford Medical Group current system guidelines.

SECONDARY OUTCOMES:
ACS Marker Evaluation | 5 years
  To evaluate early exclusion and/or inclusion of ACS with high sensitive cTn and newer cTn assays or other novel markers .

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Richard M Nowak, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States